CLINICAL TRIAL: NCT01187901
Title: Genetic Events Leading to APC-Dependent Colon Cancer in High-Risk Families; a Clinical Trial of COX and EGFR Inhibition in Familial Polyposis Patients
Brief Title: A Clinical Trial of COX and EGFR Inhibition in Familial Polyposis Patients
Acronym: FAPEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jewel Samadder, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 00039278; P01CA073992 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-24 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-05

CONDITIONS: Adenomatous Polyposis Coli
Keywords: Familial Adenomatous Polyposis; Attenuated Familial Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Erlotinib Hydrochloride; Sulindac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib and Sulindac (Active Comparator): Erlotinib 75 mg per day in combination with sulindac 150 mg twice daily for 6 months.
  Interventions: Drug: Erlotinib; Drug: Sulindac
- Placebo A and Placebo B (Placebo Comparator): Placebo capsules matching erlotinib active comparator (Placebo A) once daily and placebo capsules matching sulindac active comparator (Placebo B) twice daily for 6 months
  Interventions: Drug: Placebo A; Drug: Placebo B

INTERVENTIONS:
Drug: Erlotinib — Tarceva oral tablets are conventional, immediate-release tablets containing erlotinib as the hydrochloride salt. Erlotinib(75mg)will be taken once daily for six months in combination with sulindac.
  Other Names: Tarceva (NDA#021743)
  Arms: Erlotinib and Sulindac
Drug: Sulindac — Sulindac is a non-steroidal, anti-inflammatory indene derivative designed for the treatment of arthritic conditions. For this study, sulindac (150mg) will be taken twice daily in combination with erlotinib
  Other Names: Sulindac (ANDA#071891)
  Arms: Erlotinib and Sulindac
Drug: Placebo A — Erlotinib (Tarceva) will provide a 25 mg identical placebo. This will be provided by the Division of Cancer Prevention at the NIH who will receive the drug and placebo from the manufacturer, OSI/Genentech. Dosage for Placebo A will be 75 mg a day for 6 months.
  Other Names: Erlotinib placebo
  Arms: Placebo A and Placebo B
Drug: Placebo B — Sulindac will be encapsulated in 150 mg doses along with an identical encapsulated Placebo B. One 150 mg capsules of Placebo B will be taken twice per day with meals (breakfast and supper).
  Other Names: Sulindac placebo
  Arms: Placebo A and Placebo B

SUMMARY:
The purpose of this study is to determine in a randomized, placebo-controlled, phase II trial if the combination of sulindac and erlotinib causes a significant regression of duodenal and colorectal adenomas in familial adenomatous polyposis (FAP) and attenuated FAP (AFAP) patients.

DETAILED DESCRIPTION:
This will be a single-center, phase-II, six-month-long, placebo-controlled, double blinded, randomized trial of the epidermal growth factor receptor (EGFR) inhibitor, erlotinib (Tarceva) and the cyclooxygenase (COX-2) inhibitor, sulindac in patients with familial adenomatous polyposis (FAP) or attenuated FAP. FAP is an autosomal dominant inherited colon cancer predisposition with a 100% risk of colon cancer in the absence of preventive care (endoscopy and surgery). Efficacious chemoprevention for duodenal adenomas is an unmet clinical need in FAP patients that would reduce the morbidity from duodenectomy and risk of duodenal adenocarcinoma. Currently the only Food and Drug Administration (FDA)-approved chemopreventive agent is celecoxib which results in a modest reduction of duodenal and colorectal polyps and is associated with cardiac toxicity at effective doses. If it can be shown that combinatorial inhibition of COX-2 and EGFR activity leads to successful regression in duodenal adenomatous polyps in FAP, it could be used as an effective chemopreventive regimen in FAP patients with duodenal adenomas or who have undergone surgical resection of duodenal adenomas or have many rectal adenomas. FAP and AFAP patients will be screened by endoscopy for presence of 5 or more duodenal polyps, then randomized to either A) erlotinib at 75 mg/day and sulindac at 150 mg/day or B) placebo for 6 months. The endpoint will be endoscopy at 6 months.

Primary Aim : To determine if the combination of sulindac and erlotinib causes a significant regression of duodenal polyp burden at 6 mohths in FAP and attenuated FAP patients.

Secondary Aim: To measure if combination of sulindac and erlotinib cause a reduction in total duodenal polyp count, and change in duodenal polyp burden or count stratified by genotype and initial polyp burden.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years or older with a clinical or genetic diagnosis of FAP or attenuated FAP.
* Presence of duodenal polyps with a sum of diameters ≥ 5mm.
* Minimum of two weeks since any major surgery
* WHO performance status ≤1
* Adequate bone marrow function as show by: normal leukocyte count, platelet count ≥ 120 x 109/L, Hgb > 12 g/dL
* Adequate liver function as shown by: normal serum bilirubin(≤ 1.5 Upper Limit Normal {ULN}) and serum transaminases (≤ 2.0 ULN)
* Patient must discontinue taking any Nonsteroidal anti-inflammatory drugs (NSAIDS) within one month of treatment initiation.
* Patients must be able to provide written informed consent.

Exclusion Criteria:

* Prior treatment with any investigational drug within the preceding 4 weeks.
* Malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skins.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study as determined by the Principal Investigator such as:

  1. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia
  2. Severely impaired lung function
  3. Any active (acute or chronic) or uncontrolled infection/ disorders.
  4. Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
  5. Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Screening clinical laboratory values that indicate any of the following:

  1. anemia
  2. thrombocytopenia
  3. leucopenia
  4. elevations of transaminases greater than 2X ULN
  5. elevation of bilirubin > 1.5 X ULN
  6. alkaline phosphatase elevation > 1.5 X ULN
  7. increased creatinine, urinary protein, or urinary casts outside the clinically normal range.
* Gastrointestinal bleeding (symptoms including dyspnea, fatigue, angina, weakness, malaise, melena, hematochezia, hematemesis, anemia or abdominal pain will require clinical assessment to rule out gastrointestinal bleeding).
* Patient who is currently taking any anti-coagulation medication.
* Women who are pregnant or breast feeding.
* Patients with a known hypersensitivity to sulindac or erlotinib or to their excipients

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Burt, MD, Study Chair — University of Utah at Huntsman Cancer Institute; Niloy J Samadder, MD, Principal Investigator — University of Utah at Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sample DC, Samadder NJ, Pappas LM, Boucher KM, Samowitz WS, Berry T, Westover M, Nathan D, Kanth P, Byrne KR, Burt RW, Neklason DW. Variables affecting penetrance of gastric and duodenal phenotype in familial adenomatous polyposis patients. BMC Gastroenterol. 2018 Jul 16;18(1):115. doi: 10.1186/s12876-018-0841-8. PMID 30012100
- [Derived] Samadder NJ, Kuwada SK, Boucher KM, Byrne K, Kanth P, Samowitz W, Jones D, Tavtigian SV, Westover M, Berry T, Jasperson K, Pappas L, Smith L, Sample D, Burt RW, Neklason DW. Association of Sulindac and Erlotinib vs Placebo With Colorectal Neoplasia in Familial Adenomatous Polyposis: Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2018 May 1;4(5):671-677. doi: 10.1001/jamaoncol.2017.5431. PMID 29423501
- [Derived] Samadder NJ, Neklason DW, Boucher KM, Byrne KR, Kanth P, Samowitz W, Jones D, Tavtigian SV, Done MW, Berry T, Jasperson K, Pappas L, Smith L, Sample D, Davis R, Topham MK, Lynch P, Strait E, McKinnon W, Burt RW, Kuwada SK. Effect of Sulindac and Erlotinib vs Placebo on Duodenal Neoplasia in Familial Adenomatous Polyposis: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1266-75. doi: 10.1001/jama.2016.2522. PMID 27002448

RESULTS

PARTICIPANT FLOW:
Groups:
- Sulindac-erlotinib: Sulindac 150 mg twice daily in combination with erlotinib 75 mg per day for 6 months
- Placebo: Placebo capsules matching erlotinib active comparator (Placebo A) once daily and placebo capsules matching sulindac active comparator (Placebo B) twice daily for 6 months
Period: Overall Study
Arm/Group | Sulindac-erlotinib | Placebo
Started | 46 | 46
Completed | 37 | 36
Not Completed | 9 | 10
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Unrelated Health Reasons | 1 | 2
Not completed — Suspected Allergic Reaction | 1 | 1
Not completed — Adverse Event | 3 | 0
Not completed — No Endpoint due to Early Study Halt | 2 | 3
Not completed — Pregnancy | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sulindac-erlotinib | Placebo | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14) | 41 (14) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 18 | 18 | 36
Familial Adenomatous Polyposis (FAP) Status [Number; unit: participants]
  Classic FAP | 32 | 32 | 64
  Attenuated FAP | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Duodenal Polyp Burden From Baseline to 6 Months
Description: A comparison between the Sulindac-erlotinib and Placebo arms of the change in polyp burden from a 10-centimeter segment of the duodenum, measured as the sum of the diameters of the polyps, in millimeters (mm), from the duodenal segment (6-month polyp burden minus baseline polyp burden).
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Sulindac-erlotinib | Placebo
Number analyzed (Participants) | 46 | 46
mm | -8.5 [-9.5 to -7.0] | 8.0 [5.0 to 9.5]
Statistical Analysis 1: Comparison: Sulindac-erlotinib; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Duodenal Polyp Burden From Baseline to 6 Months in Classic Familial Adenomatous Polyposis (FAP) Participants
Description: A comparison between the Sulindac-erlotinib and Placebo arm Classic FAP subgroups of the change in polyp burden from a 10-centimeter segment of the duodenum, measured as the sum of the diameters of the polyps, in millimeters (mm), from the duodenal segment (6-month polyp burden minus baseline polyp burden).
Time Frame: Baseline and 6 months
Population: Classic FAP participants are defined as those presenting with more than 100 colonic adenomas and either (1) multiple family members with a classic FAP phenotype or (2) an adenomatous polyposis coli (APC) mutation in a region of the gene known to correlate with Classic FAP, or (3) both.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Sulindac-erlotinib | Placebo
Number analyzed (Participants) | 32 | 32
mm | -8.5 [-9.5 to -7.3] | 8.5 [4.5 to 11.3]
Statistical Analysis 1: Comparison: Sulindac-erlotinib vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in Duodenal Polyp Burden From Baseline to 6 Months in Attenuated FAP Participants
Description: A comparison between the Sulindac-erlotinib and Placebo arm Attenuated FAP subgroups of the change in polyp burden from a 10-centimeter segment of the duodenum, measured as the sum of the diameters of the polyps, in millimeters (mm), from the duodenal segment (6-month polyp burden minus baseline polyp burden).
Time Frame: Baseline and 6 months
Population: Attenuated FAP participants are defined with the presence of a mutation in a portion of the adenomatous polyposis coli (APC) gene known to correlate with attenuated FAP and presentation of a milder phenotype in terms of polyp density in the participant and the family. All participants with attenuated FAP had a confirmed mutation in the APC gene.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Sulindac-erlotinib | Placebo
Number analyzed (Participants) | 14 | 14
mm | -8.0 [-9.5 to -5.5] | 7.0 [5.0 to 9.5]
Statistical Analysis 1: Comparison: Sulindac-erlotinib vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Number of Duodenal Polyps From Baseline to 6 Months
Description: A comparison between the Sulindac-erlotinib and Placebo arms of the change in number of polyps in a 10-centimeter segment of the duodenum (6-month polyp count minus baseline polyp count).
Time Frame: Baseline and 6 months
Measure: Median (Inter-Quartile Range); unit: polyps
Arm/Group | Sulindac-erlotinib | Placebo
Number analyzed (Participants) | 46 | 46
polyps | -2.8 [-4.0 to -1.5] | 4.3 [3.1 to 5.5]
Statistical Analysis 1: Comparison: Sulindac-erlotinib vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Number of Duodenal Polyps From Baseline to 6 Months in Classic FAP Participants
Description: A comparison between the Sulindac-erlotinib and Placebo arm Classic FAP subgroups of the change in number of polyps in a 10-centimeter segment of the duodenum (6-month polyp count minus baseline polyp count)
Time Frame: Baseline and 6 months
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: polyps
Arm/Group | Sulindac-erlotinib | Placebo
Number analyzed (Participants) | 32 | 32
polyps | -2.1 [-4.0 to -0.5] | 4.0 [2.5 to 5.6]
Statistical Analysis 1: Comparison: Sulindac-erlotinib vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Number of Duodenal Polyps From Baseline to 6 Months in Attenuated FAP Participants
Description: A comparison between the Sulindac-erlotinib and Placebo arm Attenuated FAP subgroups of the change in number of polyps in a 10-centimeter segment of the duodenum (6-month polyp count minus baseline polyp count)
Time Frame: Baseline and 6 months
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: polyps
Arm/Group | Sulindac-erlotinib | Placebo
Number analyzed (Participants) | 14 | 14
polyps | -4.3 [-6.0 to -2.5] | 4.9 [3.6 to 6.0]
Statistical Analysis 1: Comparison: Sulindac-erlotinib vs Placebo; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Sulindac-erlotinib | Placebo
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 43/46 | 33/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sulindac-erlotinib (N=46) | Placebo (N=46)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 40 | 9
Oral Mucositis (Gastrointestinal disorders) | 18 | 5
Diarrhea (Gastrointestinal disorders) | 12 | 6
Nausea (Gastrointestinal disorders) | 11 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 | 10
Dry Skin (Skin and subcutaneous tissue disorders) | 7 | 7
Abdominal Pain (Gastrointestinal disorders) | 4 | 8
Dry Eye (Eye disorders) | 9 | 1
Headache (Nervous system disorders) | 4 | 8
Fatigue (General disorders) | 5 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2
Aminotransferase Increase (Investigations) | 3 | 4
Hypertension (Vascular disorders) | 3 | 0
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No